CLINICAL TRIAL: NCT04703257
Title: Evaluation of the Added Value of Metamizole to Standard Postoperative Treatment After Ambulant Shoulder Surgery: a Double-blind, Randomized Controlled Trial
Brief Title: Evaluation of the Added Value of Metamizole to Standard Postoperative Treatment After Ambulant Shoulder Surgery
Acronym: Metamizole003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jessa Hospital (Other)
Responsible Party: Principal Investigator, Stessel Björn, Dr, Principal Investigator, Jessa Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Jessa_20.91
Record Dates: First submitted 2021-01-08; First posted 2021-01-11 (Actual); Last update posted 2023-01-06 (Actual); Status verified 2023-01

CONDITIONS: Postoperative Pain; Analgesia; Surgery
Keywords: ambulant shoulder surgery; post-operative pain; recovery
MeSH Terms: conditions — Pain, Postoperative; Agnosia | interventions — Dipyrone

STUDY DESIGN:
Intervention Model Description: A monocenter, prospective, double-blind, randomized controlled superiority trial is designed to investigate the superiority of the combination of metamizole and paracetamol compared to paracetamol treatment in patients undergoing arthroscopic shoulder surgery with tendon repair.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Placebo Comparator): Patients in the control group will be instructed to take a placebo tablet three times a day for four days and patients will be instructed to take 1000 mg paracetamol orally four times a day for four days.
  Interventions: Drug: Placebo
- Intervention group (Active Comparator): Patients in the experimental group will be instructed to take metamizole 1000 mg orally three times a day for four days patients will be instructed to take 1000 mg paracetamol orally four times a day for four days.
  Interventions: Drug: Metamizole

INTERVENTIONS:
Drug: Metamizole — Patients in the experimental group will be instructed to take metamizole 1000 mg orally three times a day for four days patients will be instructed to take 1000 mg paracetamol orally four times a day for four days. .
  Arms: Intervention group
Drug: Placebo — Patients in the control group will be instructed to take a placebo tablet three times a day for four days and patients will be instructed to take 1000 mg paracetamol orally four times a day for four days.
  Arms: Control group

SUMMARY:
This study aims to investigate if the combination of metamizole and paracetamol is superior in reducing post-operative pain on day 1 after ambulatory shoulder surgery where the use of NSAIDs is prohibited compared to paracetamol treatment.

Therefore, a monocenter, prospective, double-blind, randomized controlled superiority trial will be designed to investigate the superiority of the combination of metamizole and paracetamol compared to paracetamol treatment in patients undergoing arthroscopic shoulder surgery with tendon repair.

DETAILED DESCRIPTION:
In an ambulatory setting, good post-operative analgesia is challenging because patients have to control pain at home by themselves, in the absence of hospital staff. Moreover, there is a limit in the type of analgesia that is available (i.e. no strong opioids) as well as in the route of administration (i.e. no epidural, intravenous, subcutaneous, or intramuscular route) at home. Nowadays a multimodal approach based on a combination of paracetamol, non-steroidal anti-inflammatory drugs (NSAIDs) and, if necessary, weak opioids to control pain has been advocated in the ambulatory setting. Local and regional anesthesia also has been advocated in the ambulatory setting to relieve pain for 8 to 24 hours after surgery. Despite this multimodal pain therapy, the prevalence of outpatients suffering from moderate to severe acute postoperative pain at home remains high and varies from 9 to 40%. More specifically, some patients seem to be at high risk to develop moderate to severe pain on the fourth postoperative day, among which patients undergoing arthroscopic shoulder surgery.

Besides this high prevalence, recent findings suggest that the use of NSAIDs is detrimental to tendon healing, especially in early stages. This negative impact is due to its effect on both proliferation and migration of tendon cells, as well as the inflammation reaction involved in the healing process and the bone growth necessary for tendon-to-bone healing. Healing of injured tendon proceeds through three phases: inflammation, regeneration, and remodeling/maturation. The initial phase involves an inflammatory response, in which the pro-inflammatory cyclooxygenase-2 (COX-2)/prostaglandin E2 (PGE-2) pathway is of major importance. In the regenerative phase of a tendon injury, tendon cells migrate towards a repair site, proliferate and deposit extracellular matrix (ECM) in the tissue. The expression of paxillin, a positive regulator of cell mobility, is downregulated by ibuprofen, resulting in inhibited tendon cell migration. Moreover, treatment decreases DNA synthesis and gene expression in tendon cells, harming proliferation, and interfering with normal processes of ECM remodeling. Furthermore, the resulting p21CYP1 expression and decreased Rb protein phosphorylation are associated with inhibited proliferation. Additionally, the inhibition of COX-enzymes associated with PGE-2 inhibition may lead to impaired osteoblast differentiation, essential for tendon-to-bone healing.

On top of that, NSAIDs are not always sufficiently effective, can have numerous contraindications, and are therefore not suitable in up to 25% of all patients. These controversies implicate the need for alternative pain therapy. Metamizole (dipyrone) is a non-opioid compound with strong analgesic, antipyretic, and spasmolytic effects. The analgesic efficacy of intravenous or intramuscular metamizole for pain relief after inpatient surgery is well described. Recently, we showed in a prospective, double-blind, randomized controlled trial that the combination of paracetamol and metamizole is equally effective in the treatment of acute postoperative pain at home after ambulatory surgery compared to paracetamol and ibuprofen. Moreover, patient satisfaction was equal in both groups, as well as the reported side effects.

Multiple mechanisms are involved in the antinociceptive effects of metamizole. More particularly, the inhibition of COX-1 and -2 enzymes and the activation of the endocannabinoid and opioidergic system. This seems partly similar to the working mechanism of NSAIDs, suggesting a theoretical presumption that metamizole also harms tendon repair. However, metamizole is not classified as an NSAID and no detrimental effect of metamizole on tendon healing and no link between metamizole and the previously described mechanism has been reported in the literature. The most important advantage of metamizole compared with NSAIDs is its favorable gastro-intestinal and cardiovascular side effect profile. Therefore, replacing NSAIDs with metamizole in the standard approach in surgeries where NSAIDs are contraindicated such as shoulder arthroscopies with tendon repair may increase the overall suitability of postoperative pain therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 75 years
* ASA classification 1, 2 or 3
* Bodyweight > 50 kg
* Undergoing ambulatory arthroscopic shoulder surgery and with a contraindication to NSAID (SAD ± ACJ excision or decompression, decompression + biceps tenodesis, SLAP repair, Bankart repair, rotator cuff repair)

Exclusion Criteria:

* Not meeting inclusion criteria
* Cognitive impairment or no understanding of the Dutch language
* Preoperative pharmacological pain treatment and/or a history of chronic pain excluding shoulder pain
* Allergy to or contraindication for taking the study medication (e.g. paracetamol or metamizole)
* Porphyria
* Pregnancy or lactation
* A history of severe renal, hepatic, pulmonary or cardiac failure
* A history of substance abuse, or use of medication with a suppressive effect on the central nervous system
* Hypotension
* Hematological disease
* Use of anti-rheumatic drugs
* Rhinosinusitis or nasal polyposis
* Glucose-6-phosphate dehydrogenase deficiency
* Fever or other signs of infection
* Refusal of an interscalene block

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Actual)
Dates: Start 2021-02-26 (Actual); Primary Completion 2022-12-21 (Actual); Study Completion 2022-12-21 (Actual)

PRIMARY OUTCOMES:
Postoperative pain at movement | 24 hours after the surgery
  Postoperative pain intensity at movement measured by an 11-point Numeric Rating Scale (NRS), where 0: no pain and 10: worst imaginary pain, on postoperative day 1.

SECONDARY OUTCOMES:
Quality of recovery | at baseline and days 7, 14, 28 and 3 months postoperatively
  Quality of Recovery measured by the 1-item Global Surgical Recovery (GSR) index which represents a single question about the extent to which patients consider themselves to be recovered from surgery (0-100%) at baseline and days 7, 14, 28 and 3 months postoperatively.
Quality of Recovery | at baseline and days 7, 14, 28 and 3 months postoperatively
  Measured with the EuroQol (EQ5D) questionnaire, which is non-disease specific instrument developed for describing and valuing health-related quality of life, at baseline and days 7, 14, 28 and 3 months postoperatively
Postoperative pain | at baseline, at discharge, and day 1, 2, 3, 4, 7, 14, 28, and 3 months postoperatively.
  Postoperative pain intensity at rest and at movement measured by an 11-point Numeric Rating Scale (NRS) where 0:
  no pain and 10: worst imaginary pain) at baseline, at discharge and at day 1, 2, 3, 4, 7, 14, 28 and at 3 months.
Simple shoulder test | at baseline and days 7, 14, 28, and 3 months postoperatively.
  Simple shoulder test (SST) measured at baseline and days 7, 14, 28 and 3 months postoperatively.
Adherence | day 1, 2, 3 and 4 postoperatively
  Adherence to studymedication on day 1, 2, 3 and 4 postoperatively
Adverse effects | throughout study completion, e.g. 3 months postoperatively
  Adverse effects of the studymedication
Piritramide | after surgery until discharge of PACU (up to 3 hours after surgery)
  The total amount of piritramide used in the PACU
Rescue medication | on day 1, 2, 3 and 4 postoperatively
  The use of rescue medication (tramadol) at home on day 1, 2 ,3 and 4 postoperatively (yes/no)
Satisfaction of the patient | at day 7 and 3 months postoperatively
  Satisfaction with study medication, surgery and hospital care and telephone follow-up measured at day 7 and 3 months postoperative measured by an 11-point Numeric Rating Scale (NRS) where 0: totally unsatisfied and 10: totally satisfied

CONTACTS AND LOCATIONS:
Locations (1):
- Anesthesiology Jessa hospital, Hasselt, Belgium

IPD SHARING:
Plan to Share IPD: No